CLINICAL TRIAL: NCT02630251
Title: A Phase I Open-Label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK2820151 in Subjects With Advanced or Recurrent Solid Tumors
Brief Title: Dose Escalation Study of GSK2820151 in Subjects With Advanced or Recurrent Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In 2017, GSK2820151 was terminated due to development of another BET Inhibitor (GSK525762) with a better understanding of the risk benefit profile.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201893
Record Dates: First submitted 2015-11-30; First posted 2015-12-15 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Neoplasms
Keywords: Cancer; Safety; GSK2820151; Dose escalation; Tolerability; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2820151 arm (Experimental): An accelerated dose escalation phase will be utilized in order to minimize sub-optimal drug exposures, followed by a conventional 3+3 dose escalation phase to achieve MTD. Initially, one subject per dose cohort will be recruited (accelerated dose escalation phase) until the first instance of a >=Grade 2 drug related toxicity or dose-limiting toxicity (DLT). Further cohorts will be recruited in blocks of three subjects (3+3 dose escalation phase). Projected dose levels are 3 mg, 6 mg, 12 mg, 20 mg, 40 mg, 60 mg, 100 mg, 150 mg, 200 mg, and 300 mg. Additional subjects may be enrolled at previously cleared dose levels in order to obtain further data for PK and/or PD analysis. Once MTD is determined, additional subjects (18 subjects total at MTD) may be enrolled to collect additional safety data.
  Interventions: Drug: GSK2820151

INTERVENTIONS:
Drug: GSK2820151 — GSK2820151 is provided as capsules containing 1 mg, 5 mg, 10 mg, 50 mg, or 100 mg of GSK2820151 as free base equivalent to be administered orally. The dosing regimen is as follows: Week 1 - once daily on days 1, 3, 4, and 5; Week 2 - once daily on days 1, 2, 3, 4, 5; and Weeks 3 and beyond - once daily continuously.

SUMMARY:
The study drug, GSK2820151, is a Bromodomain (BRD) and Extra-Terminal (BET) inhibitor arising from a distinct structural class. GSK2820151 potently inhibits tumor growth in vitro and in vivo in animal models. This first time in human (FTIH), open-label, dose escalation study is to assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of GSK2820151 in subjects with advanced or recurrent solid tumors. The objective is to determine the safety, tolerability and maximum tolerated dose (MTD) of GSK2820151 in subjects 18 years or older with advanced or recurrent solid tumors. Eligible subjects with advanced or recurrent solid tumors will be enrolled in the dosing cohorts until MTD is established. All subjects will receive study drug. Subjects may continue treatment in the study until disease progression, unacceptable toxicity, or withdrawal of consent. The duration of study will depend on recruitment rates and the timing of subjects' duration on study (withdrawal rates due to toxicity or progression). It is anticipated that approximately 30 to 50 subjects will be enrolled.

DETAILED DESCRIPTION:
GSK has decided to discontinue further development of GSK2820151 due to challenges in recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided
* Males and females 18 years old and greater
* Diagnosis of advanced or recurrent, histologically or cytologically confirmed, solid malignancy that is either metastatic or unresectable. At time of enrollment, subjects either refuse standard curative or palliative therapy, are not candidates for standard curative or palliative therapy, have a disease for which no non-investigational therapy exists, OR have progressed on prior therapy (up to three lines of prior cytotoxic agents are permitted).
* Subjects with solid tumors, with the exception of castration-resistant prostate cancer (CRPC), must demonstrate measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* All prior treatment- related toxicities must be National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 <=Grade 1 (except alopecia [permissible at any Grade] and peripheral neuropathy [which must be <= Grade 2]) at the time of treatment allocation.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1.
* Adequate organ function defined as follows: System and Laboratory Values: Hematologic - Absolute neutrophil count (ANC) >=1.5 X 10^9/liter (L), Hemoglobin >=9 grams (g)/deciliter (dL) (subjects that required transfusion or growth factor need to demonstrate stable hemoglobin for 7 days of 9 g/dL), Platelets >=100 X 10^9/L, prothrombin time (PT)/ international normalized ratio (INR) and partial thromboplastin time (PTT) - <=1.5 X upper limit of normal (ULN); Hepatic - Albumin >=2.5 g/dL, Total bilirubin <=1.5 X ULN (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35% or subject has a diagnosis of Gilbert's syndrome), Alanine aminotransferase (ALT) <=2.5 x ULN OR <5 x ULN is acceptable for subjects with documented liver metastases/tumor infiltration; Renal - Creatinine <=1.5 X ULN OR Creatinine clearance [either directly measured or calculated by Cockcroft-Gault formula] >=40 milliliter (mL)/minute (min); Cardiac - Ejection fraction >=50% by echocardiogram or multigated acquisition scan (MUGA), Troponin (T) <=ULN, Potassium >=Lower limit of normal (LLN) and <=ULN, Magnesium >=LLN
* Able to swallow and retain orally administered medication.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, or documented bilateral tubal oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 units (U)/mL and estradiol <40 picograms (pg)/mL (<140 picomoles (pmol)/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. Child-bearing potential and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 7 months after the last dose of study medication. Negative serum pregnancy test <=7 days prior to first study drug dose. Female subjects who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for 5 half-lives of GSK2820151 or at least 28 days (whichever is longer) following the last dose of study treatment.
* Male subjects with female partners of child bearing potential must agree to use one of the methods of contraception specified. This method must be used from the time of the first dose of study medication until 16 weeks after the last dose of study medication. In addition, male subjects whose partners are or become pregnant on study medication must continue to use condoms for 7 days after stopping study medication

Exclusion Criteria:

* Primary malignancy of the central nervous system or malignancies related to human immunodeficiency virus (HIV) or solid organ transplant.
* More than three prior lines of cytotoxic therapy.
* Recent prior therapy, defined as follows: 1) Any investigational or Food and Drug Administration (FDA)-approved anti-cancer drug within 14 days or 5 half-lives, whichever is longer, prior to the first dose of GSK2820151. Any nitrosoureas or mitomycin C within 42 days prior to the first dose of GSK2820151. Prior therapy with monoclonal antibodies is permitted so long as 14 days have elapsed since therapy and all therapy-related toxicity has resolved to Grade 1 or less. Note that an investigational drug is defined as a drug without an approved oncologic indication.

  2) Any radiotherapy within 14 days or major surgery within 28 days prior to the first dose of GSK2820151.

  3) Anti-androgen therapies for prostate cancer, such as bicalutamide, must be stopped 4 weeks prior to enrollment. Second-line hormone therapies such as enzalutamide, abiraterone, or orteronel should be stopped 2 weeks prior to enrolment. Subjects with prostate cancer should remain on luteinizing hormone releasing hormone (LHRH) agonists or antagonists. Subjects with prostate cancer may also remain on low-dose prednisone or prednisolone (up to 10 milligrams [mg]/day) and still be eligible for this study.

  4) In addition, any therapy-related toxicity must have resolved to Grade 1 or less, with the exception of alopecia (acceptable at any Grade) and peripheral neuropathy (which must be Grade 2 or less prior to enrollment).
* Therapeutic anticoagulation (e.g., warfarin, heparin) must be discontinued and coagulation parameters must be normalized prior to the first dose of GSK2820151. Low dose (prophylactic) low molecular weight heparin (LMWH) is permitted. In addition, INR must be monitored in accordance with local institutional practices.
* Current use of a prohibited medication or planned use of any forbidden medications during treatment with GSK2820151.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. NOTE: Subjects previously treated for these conditions that have had stable central nervous system (CNS) disease (verified with consecutive imaging studies) for >1 months, are asymptomatic and off corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to study Day 1 are permitted. Stability of brain metastases must be confirmed with imaging. Subject treated with gamma knife therapy can be enrolled 2 weeks post-procedure as long as there are no post-procedure complications/stable. In addition, subjects treated or currently taking enzyme-inducing anticonvulsant (EIAC) are allowed on study.
* Cardiac abnormalities as evidenced by any of the following: History of or current "untreated" clinically significant uncontrolled arrhythmias, Clinically significant conduction abnormalities or arrhythmias, Presence of cardiac pacemaker, History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA), History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months. Subjects with a history of stent placement requiring ongoing antithrombotic therapy (e.g., clopidogrel, prasugrel) will not be permitted to enroll.
* Any of the following electrocardiogram (ECG) findings: Baseline QTcF >=450 millisecond (msec). NOTE: Any clinically significant ECG assessments should be reviewed by the site cardiologist prior to study entry.
* Any of the following liver findings: ALT >2.5xULN, ALT > 5xULN with liver metastases/tumor infiltration, Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment). NOTE: Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, persistent jaundice or cirrhosis
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. History of known HIV infection. NOTE: Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) polymerase chain reaction (PCR) is obtained.
* Any serious known immediate or delayed hypersensitivity reaction(s) to GSK2820151 or idiosyncrasy to drugs chemically related to the investigational drug.
* Hemoptysis >1 teaspoon in 24 hours within the last 28 days.
* History of major gastrointestinal bleeding within the last 6 months.
* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-agent open-label dose escalation study to determine the Maximum tolerated dose (MTD)
Pre-assignment Details: The study was terminated due to development of another bromodomain and extra-terminal(BET) Inhibitor with a better understanding of the risk benefit profile.
Groups:
- GSK2820151 3 mg: Participants received GSK2820151 capsules at a dose of 3 milligram (mg) once daily on days 1, 3, 4 and 5 on Week 1, during Week 2 once daily on days 1, 2, 3, 4, and 5. Participants received GSK2820151 3 mg once daily from Week 3 onwards every 4 weeks, until the end of the treatment.
- GSK2820151 6 mg: Participants received GSK2820151 capsules at a dose of 6 mg once daily on days 1, 3, 4 and 5 on Week 1, during Week 2 once daily on days 1, 2, 3, 4, and 5. Participants received GSK2820151 6 mg once daily from Week 3 onwards every 4 weeks, until the end of the treatment.
- GSK2820151 12 mg: Participants received GSK2820151 capsules at a dose of 12 mg once daily on days 1, 3, 4 and 5 on Week 1, during Week 2 once daily on days 1, 2, 3, 4, and 5. Participants received GSK2820151 12 mg once daily from Week 3 onwards every 4 weeks, until the end of the treatment.
- GSK2820151 20 mg: Participants received GSK2820151 capsules at a dose of 20 mg once daily on days 1, 3, 4 and 5 on Week 1, during Week 2 once daily on days 1, 2, 3, 4, and 5. Participants received GSK2820151 20 mg once daily from Week 3 onwards every 4 weeks, until the end of the treatment.
Period: Overall Study
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Started | 2 | 1 | 1 | 1
Completed | 2 | 1 | 0 | 1
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 0 | 0 | 2
  >=65 years | 0 | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 4
  Male | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European Heritage | 2 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or suspected transmission of an infectious agent via the study drug were categorized as SAE.
Time Frame: 2 years 8 months
Population: All Treated Population included all participants who received at least one dose of GSK2820151.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants
  AEs | 2 | 1 | 1 | 1
  SAEs | 2 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Dose Delays and Reduction
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Withdrawn Due to Toxicities
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Withdrawals due to toxicities were evaluated.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Clinical Chemistry Parameters
Description: Blood samples were collected at indicated time-points for the analysis of clinical chemistry parameters like total and direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total protein, albumin, sodium, potassium, calcium, blood urea nitrogen (BUN), creatinine, chloride, fasting glucose, ionized calcium, gamma-glutamyltransferase, total carbon dioxide , uric acid, and magnesium.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Hematology Parameters
Description: Blood samples were collected at indicated time-points for the analysis of hematology parameters like hemoglobin (HGB), platelet count, red blood cell (RBC) count, white blood cell (WBC) count, neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Urinalysis Parameters
Description: Urine samples were collected at indicated time-points for the analysis of urinalysis parameters like potential of hydrogen (pH), microscopic examination, specific gravity, ketones, protein, glucose, and blood.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Gastrointestinal Parameters
Description: Blood samples were collected at indicated time-points for the analysis of gastrointestinal parameters like cytokines and C-peptide.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Vital Signs Parameters
Description: Vital signs included systolic blood pressure and diastolic blood pressure, heart rate, and temperature.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Abnormalities for Electrocardiogram (ECG)
Description: Triple 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measures PR, QRS, QT and corrected QT using Fridericia's formula (QTcF) intervals.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. DLTs included Grade 4 neutropenia, Febrile neutropenia, Grade 4 anemia, Grade 3 thrombocytopenia, Alanine aminotransferase (ALT) >3 times upper limit of normal (ULN) plus bilirubin >=2 times ULN (>35 percent direct) or ALT between 3-5 times ULN with bilirubin < 2 times ULN but with hepatitis symptoms or rash, Grade 3 nausea, vomiting or diarrhea, Grade 3 hypertension, Grade 4 hypertension, Grade 3 or greater clinically significant non-hematologic toxicity, Grade 2 troponin B elevation were considered as DLT.
Time Frame: Up to 4 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Changes in Cardiac Safety Including Corrected QT Interval (QTc)
Description: Changes in cardiac parameters like QTc, PR Interval, QRS duration, and QT interval were assessed. Baseline is defined as the most recent, non-missing value prior to or on the first study treatment dose date for GSK2820151. Change from baseline was calculated as visit value minus Baseline value.
Time Frame: Baseline and up to 2 years 8 months
Population: All Treated Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Milliseconds | -5.33 (17.272) | -9.25 (13.849) | 4.91 (11.274) | -24.95 (10.400)

12. Secondary Outcome: Changes in Cardiac Safety Including Heart Rate
Description: Change in heart rate was assessed. Baseline is defined as the most recent, non-missing value prior to or on the first study treatment dose date for GSK2820151. Change from baseline was calculated as visit value minus Baseline value.
Time Frame: Baseline and up to 2 years 8 months
Population: All Treated Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Beats per minute | -0.44 (7.719) | 11.51 (8.072) | 3.41 (5.929) | 2.03 (4.609)

13. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR is defined as the percentage of participants with a confirmed complete response (CR) or a partial response (PR) at any time as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Percentage of participants | 0 | 0 | 100 | 0

14. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the interval of time (in weeks) between the start date of treatment and the earlier of the date of disease progression and the date of death due to any cause. PFS was censored at the last adequate assessment where visit level response is CR, PR, or stable disease.
Time Frame: 2 years 8 months
Population: All Treated Population
Measure: Number; unit: Weeks
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Weeks
  Participant 1 | 5.3 | 0 | 0 | 0
  Participant 2 | 9.9 | 0 | 0 | 0
  Participant 3 | 0 | 8.4 | 0 | 0
  Participant 4 | 0 | 0 | 72.1 | 0
  Participant 5 | 0 | 0 | 0 | 8.1

15. Secondary Outcome: Protein Biomarker (Cytokines and Acute Phase Proteins) Analysis for Pharmacodynamic (PD) Data
Description: Blood samples were planned to be collected for analysis of protein PD biomarkers like cytokines and acute phase proteins.
Time Frame: 2 years 8 months
Population: PK Population. Data was not collected for this endpoint as the study was terminated.
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Messenger Ribonucleic Acid (mRNA) Analysis for PD Data
Description: Blood samples were planned to be collected for analysis of mRNA.
Time Frame: 2 years 8 months
Population: PK Population. Data was not collected for this endpoint as the study was terminated.
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of Cmax. The average Standard Deviation (SD) for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. Pharmacokinetic (PK) parameters were conducted by non-compartmental methods using Phoenix WinNonlin. PK Population consisted of all subjects from the All Treated Population for whom a PK sample is obtained and analyzed
Time Frame: Week 1, Day 1 (Pre-dose, 15 and 30 minutes, 1, 2, 4, 8, 16, 24 and 33 hours post-dose); Week 3, Day 4 (Pre-dose, 15 and 30 minutes, 1, 2, 4, 8, 16, 24 and 48 hours)
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Nanograms per milliliter | 31.78 (9.599) | 35.08 (1.061) | 36.17 (8.237) | 148.11 (14.595)

18. Secondary Outcome: Time to Cmax (Tmax) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of Tmax. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Hours | 1.50 [1.00 to 2.00] | 2.50 [1.00 to 4.00] | 1.00 [1.00 to 2.00] | 0.75 [0.5 to 1.00]

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Time (AUC[0-t]) of GSK2820151
Description: Blood samples were collected at indicated time-points for analysis of AUC(0-t). The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours* nanogram per milliliter
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Hours* nanogram per milliliter | 356.10 (237.739) | 392.17 (54.801) | 211.84 (16.349) | 958.35 (92.900)

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC[0-inf])
Description: Blood samples were collected at indicated timepoints for analysis of AUC(0-inf). The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters was conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours* nanogram per milliliter
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Hours* nanogram per milliliter | 488.40 (381.276) | 479.12 (127.755) | 216.65 (18.215) | 1107.74 (147.297)

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Tau (AUC[0-tau]) of GSK2820151
Description: Blood samples were collected at indicated time-points for analysis of AUC(0-tau). The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours* nanogram per milliliter
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Hours* nanogram per milliliter | 328.55 (209.993) | 377.60 (75.413) | 210.32 (16.761) | 918.11 (149.815)

22. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of GSK2820151
Description: Blood samples were collected at indicated time-points for analysis of t1/2. The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Hours | 11.66 (6.300) | 10.91 (1.153) | 4.77 (0.336) | 10.14 (1.379)

23. Secondary Outcome: Trough Concentration (Ctau) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of Ctau. The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Nanograms per milliliter | 7.02 (6.674) | 6.04 (2.871) | 0.91 (0.276) | 12.77 (2.036)

24. Secondary Outcome: Accumulation Ratio (Ro) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of Ro. Ro was calculated as the ratio of AUC(0-tau) on Week 3 Day 4 divided by AUC(0-tau) on Week 1 Day 1. The ratio was calculated from AUC(0-tau) on Week 3 Day 4 and AUC(0-tau) on Week 1 Day 1 parameters for each participant.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Ratio | 1.17 (0.999) | 1.33 (NA) — Standard deviation could not be derived as a single participant was analyzed | 0.95 (NA) — Standard deviation could not be derived as a single participant was analyzed | 1.26 (NA) — Standard deviation could not be derived as a single participant was analyzed

25. Secondary Outcome: Time Invariance of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of time invariance. Time invariance was calculated as the ratio of AUC(0-tau) on Week 3 Day 4 divided by AUC(0-inf) on Week 1 Day 1. The ratio for SD was calculated from AUC(0-tau) on Week 3 Day 4 and AUC(0-inf) on Week 1 Day 1 parameters for each participant.
Time Frame: as for outcome 17
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Ratio | 0.87 (0.366) | 1.10 (NA) — Standard deviation could not be derived as a single participant was analyzed | 0.92 (NA) — Standard deviation could not be derived as a single participant was analyzed | 1.02 (NA) — Standard deviation could not be derived as a single participant was analyzed

26. Secondary Outcome: Clearance (CL/F) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of CL/F. The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Liters per hour | 11.29 (8.910) | 12.96 (3.373) | 66.92 (15.339) | 18.21 (2.425)

27. Secondary Outcome: Volume of Distribution (Vz/F) of GSK2820151
Description: Blood samples were collected at indicated timepoints for analysis of Vz/F. The average SD for each participant was calculated over indicated time points Week 1, Day 1and Week 3, Day 4. PK parameters were conducted by non-compartmental methods using Phoenix WinNonlin.
Time Frame: as for outcome 17
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
Number analyzed (Participants) | 2 | 1 | 1 | 1
Liters | 136.07 (63.572) | 201.07 (31.480) | 455.65 (72.602) | 268.91 (71.679)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of study treatment up to 2 years 8 months.
Description: Non-serious AEs and SAEs were reported for the All Treated Population which comprised of all participants who received at least 1 dose of GSK2820151.
Arm/Group | GSK2820151 3 mg | GSK2820151 6 mg | GSK2820151 12 mg | GSK2820151 20 mg
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/1 | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2820151 3 mg (N=2) | GSK2820151 6 mg (N=1) | GSK2820151 12 mg (N=1) | GSK2820151 20 mg (N=1)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2820151 3 mg (N=2) | GSK2820151 6 mg (N=1) | GSK2820151 12 mg (N=1) | GSK2820151 20 mg (N=1)
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Lymphoedema (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Urine abnormality (Investigations) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemoglobin decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperaesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Flank pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Cardiac disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02630251/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02630251/SAP_001.pdf